CLINICAL TRIAL: NCT02262078
Title: Acute Effects of Inhaled Sodium Nitrite on Cardiovascular Hemodynamics in Heart Failure With Preserved Ejection Fraction
Brief Title: Inhaled Sodium Nitrite on Heart Failure With Preserved Ejection Fraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Aires Pharmaceuticals, Inc. (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Barry Borlaug, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 14-005091; R01HL128526 (NIH); U10HL110262 (NIH)
Record Dates: First submitted 2014-09-30; First posted 2014-10-10 (Estimated); Results first posted 2017-01-19 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-07

CONDITIONS: Heart Failure
Keywords: Preserved Ejection Fraction
MeSH Terms: conditions — Heart Failure | interventions — Sodium Nitrite; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Saline) (Placebo Comparator): Participants receive normal saline, administered by inhalation over 10-15 minutes, using a nebulizer
  Interventions: Other: Placebo
- Sodium Nitrite (Experimental): Participants receive Sodium Nitrite inhalation solution, administered by inhalation over 10-15 minutes, using a nebulizer
  Interventions: Drug: Sodium Nitrite Inhalation Solution

INTERVENTIONS:
Drug: Sodium Nitrite Inhalation Solution — 90mg of (nebulized) inhaled sodium nitrite will be administered (by inhalation) to participants prior to exercise.
  Other Names: AIR001, NaNO2, Sodium Nitrite
  Arms: Sodium Nitrite
Other: Placebo — Normal saline will be administered (by inhalation) to participants prior to exercise.
  Other Names: Saline
  Arms: Placebo (Saline)

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) is a major public health problem that has no proven effective treatment. This study will assess the effects of nebulized inhaled nitrite administration on resting and exercise hemodynamics in patients with HFpEF referred to the catheterization lab.

DETAILED DESCRIPTION:
Patients referred to the cardiac catheterization laboratory for invasive exercise stress testing will be prospectively recruited. Standard right heart catheterization using high fidelity micromanometers (Millar Instruments) will be performed at rest and during supine exercise with simultaneous expired gas analysis (Medgraphics) as is the investigator's current practice. The protocol is rest-passive leg elevation--20 Watts exercise x 5 minutes, and then graded workload increases in 10Watt increments (3 minute stages) to exhaustion. Hemodynamic, arterial and mixed venous blood gas and expired gas data are acquired at rest, during each exercise stage and at peak exercise. Venous blood samples will be obtained at rest and at peak exercise. Perceived symptoms of dyspnea and fatigue will be quantified using the Borg dyspnea and effort scores at each stage of exercise.

After the initial exercise study and hemodynamics have returned to baseline, previously prepared study drug (normal saline placebo or Sodium Nitrite Inhalation Solution (AIR001) 90mg placed into the medication chamber) will be nebulized utilizing the Aerogen Solo-Idehaler over 10-15 minutes. After a 15 minute observation period post completion of nebulization, resting hemodynamic and expired gas data will be acquired exactly as in the initial run. Subjects will then repeat the leg elevation-20 Watt x 5 minutes exercise phase. Blood samples will be again obtained at rest and with exercise. Subjects will repeat exercise only at the 20 Watt stage, rather repeating the entire study. This is done to increase the feasibility and shorten the time of the case. The investigators have previously observed that the vast majority (>85%) of the elevation in cardiac filling pressures and reduction in venous oxygen content in people with HFpEF occurs at the low 20 Watt workload, so repeating exercise hemodynamic assessment at this load should be sufficient to detect any clinically meaningful treatment effect.

ELIGIBILITY:
Inclusion Criteria:

* Heart Failure with preserved Ejection Fraction (HFpEF) is defined by clinical symptoms of dyspnea and fatigue
* Normal left ventricular ejection fraction (>/=50%)
* And elevated Left Ventricular (LV) filling pressure at cardiac catheterization (defined as resting Pulmonary Capillary Wedge Pressure (PCWP)>15 mmHg and/or PCWP >/=25 mmHg during exercise).

Exclusion Criteria:

* Systolic Blood Pressure <120 mmHg (during catheterization)
* Prior nitrate therapy (within previous 2 weeks)
* Glucose-6-Phosphate Dehydrogenase (G6PD) deficiency
* Other "non-HFpEF" specific causes of heart failure such as significant valvular disease (>moderate left-sided regurgitation, >mild stenosis)
* Severe pulmonary disease
* Unstable coronary disease or coronary spasm
* Primary renal or hepatic disease (end stage renal failure/on dialysis or clinical diagnosis of hepatitis or hepatic cirrhosis)
* Constrictive pericarditis, or infiltrative, restrictive, or hypertrophic cardiomyopathies
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry Borlaug, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Borlaug BA, Melenovsky V, Koepp KE. Inhaled Sodium Nitrite Improves Rest and Exercise Hemodynamics in Heart Failure With Preserved Ejection Fraction. Circ Res. 2016 Sep 16;119(7):880-6. doi: 10.1161/CIRCRESAHA.116.309184. Epub 2016 Jul 25. PMID 27458234
- [Derived] Reddy YNV, Stewart GM, Obokata M, Koepp KE, Borlaug BA. Peripheral and pulmonary effects of inorganic nitrite during exercise in heart failure with preserved ejection fraction. Eur J Heart Fail. 2021 May;23(5):814-823. doi: 10.1002/ejhf.2093. Epub 2021 Feb 1. PMID 33421267

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were referred to the Rochester, Minnesota Mayo Clinic cardiac catheterization laboratory for invasive hemodynamic exercise stress testing between December 2014 and December 2015.
Pre-assignment Details: Of 70 patients screened, 32 were excluded based upon entry criteria and 12 were excluded based on hemodynamic criteria for Heart Failure with preserved Ejection Fraction (HFpEF) (n=10) or because arterial pressures were too low (n=2).
Period: Overall Study
Arm/Group | Placebo (Saline) | Sodium Nitrite
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Saline) | Sodium Nitrite | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (10) | 67 (9) | 70 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 5 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 13 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Pulmonary Capillary Wedge Pressure During Exercise
Description: Pulmonary capillary wedge pressure is a measure of cardiac filling pressure, measured in millimeters of mercury (mmHg)
Time Frame: Baseline, after study drug dosing, approximately 4 minutes after starting exercise
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Placebo (Saline) | Sodium Nitrite
Number analyzed (Participants) | 13 | 13
millimeters of mercury | -1 (2) | -4 (3)
Statistical Analysis 1: Comparison: Placebo (Saline) vs Sodium Nitrite; Test type: Superiority or Other; p = 0.002, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From baseline to X hours following treatment.
Arm/Group | Placebo (Saline) | Sodium Nitrite
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 1/13 | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Saline) (N=13) | Sodium Nitrite (N=13)
Vasovagal syncope (Cardiac disorders) | 1 (1) | 0 (0) — One episode of vasovagal syncope 4 hours after completing study
Taste perversion (General disorders) | 0 (0) | 1 (1) — Salty taste following the nebulizer treatment

LIMITATIONS AND CAVEATS:
Patients with symptoms that might independently cause symptoms were excluded, including severe valvular or coronary heart disease and advanced lung, liver or kidney disease. Cannot determine if results would apply to these co-morbidities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes